CLINICAL TRIAL: NCT06621511
Title: OurSleepKit: A Couple-focused m-Health Intervention to Support Adherence to CPAP Treatment
Brief Title: OurSleepKit To Support CPAP Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB #: 24-04-26; R01HL160836 (NIH)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; CPAP Treatment; Treatment Adherence
Keywords: Obstructive Sleep Apnea; CPAP Treatment; Mobile Health; Treatment Adherence; Dyadic Coping; Couple
MeSH Terms: conditions — Sleep Apnea, Obstructive; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Couples in the intervention group will have exposure to the OurSleepKit app in addition to usual care.
- Control group (No Intervention): Couples in the control group will not have exposure to the OurSleepKit app during the trial. Patients will receive usual care.

INTERVENTIONS:
Behavioral: OurSleepKit — OurSleepKit is developed as an app including a patient version and a partner version, to be downloaded on the patient's or partner's mobile devices at home. The goal of OurSleepKit is to coach mutual engagement and model positive partner involvement in CPAP treatment, thus motivating greater CPAP adherence. Using OurSleepKit, both the patient and partner will complete periodic assessments tracking various aspects of their sleep and CPAP use. The assessment data are then processed by OurSleepKit to provide customized and dynamically updated support content consisting of brief story-telling videos featuring real-life couples' experiences emphasizing positive dyadic coping and problem-solving strategies. OurSleepKit delivers timely tailored prompts through push notifications on the users' mobile devices' screens, linked to relevant support content, to facilitate positive conversation in the dyad and offer in-the-moment support for CPAP use.

SUMMARY:
The goal of this clinical trial is to learn if a couple-focused mobile health intervention will improve the use of continuous positive airway pressure (CPAP), the primary treatment option for obstructive sleep apnea (OSA). Participants include newly diagnosed patients with OSA who are candidates for CPAP treatment and their partners. The couples will received supportive information and resources on their mobile devices before CPAP begins and continuing for 6 months into CPAP treatment. Their interaction with the resources is self-paced and the time sent engaging with the information is up to them. Participants will be asked to answer questions independently at five points: before CPAP, and after using CPAP for 1-week, 1-month, 3-months and 6-months. Those questions are about their experience of using CPAP, how the partner is involved in CPAP treatment, and symptoms and quality of life. At the end of the study, some couples may be contacted for a virtual discussion about your experience regarding study participation which lasts approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* patients should be males or females (age≥18 years) with diagnosed OSA and candidates for CPAP therapy (with any type of pressure delivery mode), and are cohabiting with their partner for at least one year
* The partners of eligible patients will be recruited if they are not diagnosed with OSA and not using CPAP
* both partners should have their own mobile devices with access to the internet

Exclusion Criteria:

* have a diagnosis of a sleep disorder other than OSA based on a polysomnogram (e.g., central sleep apnea, narcolepsy, or periodic limb movement disorder)
* have planned bariatric surgery (as they typically quit CPAP after surgery)
* have a partner using CPAP
* are pregnant because the changes in respiration and sleep quality occurring with pregnancy may confound the results.
* couples with one or both partners doing regular overnight shift work or those unable to speak or write in English will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
CPAP adherence | 6 months
  Average hours of nightly CPAP use over the course of the first six months of treatment

SECONDARY OUTCOMES:
Self-efficacy | 6 months
  Self-Efficacy Measure for Sleep Apnea (SEMSA) is a 26-item validated instrument that contains 3 subscales: risk perception of OSA, outcome expectancies of CPAP, and treatment self-efficacy. Internal consistency was reported as 0.90 for the total scale and 0.85 to 0.89 for the 3 subscales. Reported test-retested reliabilities ranged from 0.68 to 0.77.96
Functional Status | 6 months
  Functional Outcomes of Sleep Questionnaire (FOSQ) is a 30-item disease-specific measure to assess the impact of excessive daytime sleepiness on activities of daily living. It includes five subscales: activity level, vigilance, intimacy and sexual relationships, general productivity, and social outcomes. The potential range for each subscale is 1-4, with a total score of 5-20. Higher scores on the FOSQ indicate better daily functioning. The FOSQ has established content validity, test-retest reliability (0.90), internal consistency (0.96), and concurrent validity with standardized generic measures of functional status.
Health-Related Quality of life | 6 months
  Quality of life will be measured by the 12-item Short Form Health Survey (SF-12). The SF-12 is a validated short form survey with 12 questions selected from the SF-36 Health Survey. The questions are scored to provide evaluations into mental and physical functioning and overall health-related quality of life.
Dyadic Coping | 6 months
  The Dyadic Coping Inventory (DCI) is a 37-item questionnaire that assesses stress communication and dyadic coping as perceived by each partner about his or her own coping, each partner's perception of the other's coping, and each partner's view of how they cope as a couple on a scale from 1 (very rarely) to 5 (very often). There are four subscales measuring types of dyadic coping: delegated, supportive, stress communication, and negative dyadic coping.
Daytime Sleepiness | 6 months
  Epworth Sleepiness Scale (ESS) includes items about the likelihood of falling asleep in eight soporific situations. The ESS significantly correlates with the frequency of apneic episodes and is a clinical and research standard in the assessment of daytime sleepiness. It has high test-retest reliability (0.82) and internal consistency (0.88).
Sleep Quality and Sleep-related Impairment | 6 months
  Patient-Reported Outcomes Information System (PROMIS®) assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep.The PROMIS Sleep-Related Impairment focuses on self- reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Both tools can readily discriminate patient and control groups, and are sensitive to treatment.
Partner Involvement in CPAP Treatment | 6 months
  A brief questionnaire with 6 validated items will be used, including three subscales: pressure (asked about using CPAP, tried to persuade you to use CPAP, dropped hints about using CPAP), collaboration (helped solve a problem with CPAP, helped with the CPAP machine), and support (felt supported for using CPAP) on a scale from 1 (not at all) to 5 (extreme). We have used paired versions (one for patient and one for partner) for dyadic evaluation.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northeastern University, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be shared per NIH policy after the completion and publication of the main analyses. The final research data will not contain any patient identifiers.
Supporting Information: Study Protocol, ICF